CLINICAL TRIAL: NCT03764202
Title: Determination of Sufentanil in Breast Milk of Puerpera During Analgesia
Brief Title: Determination of Sufentanil in Breast Milk of Puerpera
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WUWQNXM 2015-1-36
Record Dates: First submitted 2018-11-25; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Cesarean Section

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CSEA，1μg/kg•d (Other): * The puerpera received combined spinal epidural anesthesia
  * The dosage of sufentanil intravenous analgesia was 1 μg/kg•d
  Interventions: Other: Detection of sufentanil concentration
- CSEA，1.5μg/kg•d (Other): * The puerpera received combined spinal epidural anesthesia
  * The dosage of sufentanil intravenous analgesia was 1.5 μg/kg•d
  Interventions: Other: Detection of sufentanil concentration
- GA，1μg/kg•d (Other): * The puerpera received general anesthesia
  * The dosage of sufentanil intravenous analgesia was 1 μg/kg•d
  Interventions: Other: Detection of sufentanil concentration
- GA，1.5μg/kg•d (Other): * The puerpera received general anesthesia
  * The dosage of sufentanil intravenous analgesia was 1.5 μg/kg•d
  Interventions: Other: Detection of sufentanil concentration
- CSEA，Epidural analgesia (Other): * The puerpera received combined spinal epidural anesthesia
  * Postoperative analgesia was performed with epidural analgesia
  * Speed of epidural analgesia pump ：6ml/h（0.1% ropivacaine , 0.5μg/ml sufentanil）
  Interventions: Other: Detection of sufentanil concentration

INTERVENTIONS:
Other: Detection of sufentanil concentration — * Concentration of sufentanil in human breast milk was determined by LC-MS /MS method
  * The volume of human breast milk was detected at each fixed time point

SUMMARY:
To determination of sufentanil in human breast milk during the administration of the sufentanil via the analgesic infusion pump and after the administration, to determine whether the breastfeeding after clinical anesthetic or analgesic administration has an effect on the infant and provide a reference for the security issues.

DETAILED DESCRIPTION:
The concentration of sufentanil in milk was determined by LC-MS /MS method( liquid chromatography mass spectrometry).The separation was carried on Agilent ZORBAX Eclipse Plus C18 column(2.1×50 mm, 3.5 μm)with a mobile phase of 10 mmol ammonium formate(A)and methanol(B), and the elution conditions were optimized as follows：linear gradient 0→0.30 min, A:B=50:50; 0.30→0.31 min, A:B=50:50→10:90; 3.00→3.10 min, A:B=10:90→50:50; 3.1→6.5min, A:B=50:50; The flowing rate was 0.2 mL•min-1, column temperature was 30 ℃, injection volume was 5 μL. ESI source was applied and operated in positive ion mode. Quantitative determination was performed using multiple reaction monitoring (MRM) of m/z 387.2 → m/z 238.2 for sufentanil, and m/z 337.2 → m/z 158.2 for fentanyl.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20yr to 38yr
* Height 155~170 cm
* Weight 65~85 Kg
* American Society of Anesthesiologists statuses I or II
* Normal cardiac and pulmonary function
* Undergoing elective Cesarean section
* Willing to provide breast milk

Exclusion Criteria:

* pregnancy induced hypertension
* gestational diabetes
* gestational heart disease

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The concentration of sufentanil in human breast milk | 1 year
  The concentration of sufentanil in human breast milk was detected at each fixed time point
The volume of human breast milk | 1 year
  The volume of human breast milk was detected at each fixed time point
The dose of sufentanil in human breast milk | 1 year
  The amount of sufentanil in the milk multiplied by the concentration of sufentanil and the volume of milk at each fixed time point

CONTACTS AND LOCATIONS:
Overall Officials: Zhang liangcheng, M.D., Principal Investigator — Fujian Medical University Union Hospital